CLINICAL TRIAL: NCT00498498
Title: A Multicenter Observational Study to Evaluate Dynamics of Endothelin and Markers of Cellular Apoptosis in Cerebrospinal Fluid and Plasma in Moderate and Severe Human Head Injury
Brief Title: Observational Endothelin and Markers of Cellular Apoptosis In CSF Head Injury
Acronym: Endothelin
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: S001.2; S001; S001.1; S001.2
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Cerebrovascular Trauma; Neurohormones; Cellular Apoptosis; Endothelin System
Keywords: severe head injury; Endothelin; CSF; Plasma; Cellular Apoptosis
MeSH Terms: conditions — Cerebrovascular Trauma; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF, plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to answer the following questions:

* What is the time course of the expected changes in endothelin levels during the first two weeks after injury and how does this relate to outcome?
* What is the relation between endothelin levels (big ET-1 and ET-1) in plasma and cerebrospinal fluid and type of injury, from CT scans and GCS?
* What is the relation between endothelin levels (big ET-1 and ET-1) in plasma and cerebrospinal fluid and outcome measurements like GOSE, ICP and CT scans?
* What is the relation between neurohormones related to the neutral endopeptidase (NEP) (ANP, BNP and cGMP) in plasma and cerebrospinal fluid and type of injury, from CT scans and GCS?
* What is the relation between endothelin levels (big ET-1 and ET-1) in plasma and cerebrospinal fluid and markers for apoptosis?

DETAILED DESCRIPTION:
Severe traumatic brain injury (TBI) remains a critical problem in the United States and throughout the world. Advances in critical care of the TBI patient has resulted in improved outcome. However, despite these efforts, half of the patients with severe brain injury die or are left with severe disability. Thus, the need for a pharmaceutical agent to blunt the cascade of neurotoxins released with mechanical head trauma and improve outcome is critically important. One of these neurotoxins is endothelin, a potent vasoactive peptide, which is considered to play a major role in TBI, particularly with subarachnoid hemorrhage and concomitant vasospasm. However, relatively little is known regarding the up-regulation of this toxin after head injury. Thus, the purpose of this observational study is to document the levels of endothelin in cerebrospinal fluid and plasma of patients with brain injury over a 14 day period. Aliquots of CSF and blood will be obtained at 12 hour intervals as long as a ventriculostomy for sampling of CSF is required for routine management. Additional information regarding the severity of injury, CT pathology, intracranial pressure, neurologic assessment, CSF biomarkers, and transcranial doppler ultrasound will also be collected. The study will be implemented among 12 centers,8 in the U.S.A and 3 in Europe and 1 in Canada, providing an average of approximately 5 patients per center over a period of 7 months. The study may be extended based on an interim analysis of endothelin levels at various injury severity levels. Data will be collected and coordinated by the American Brain Injury Consortium utilizing a web-based entry system. Following the completion of accrual a final report will be assembled by the ABIC which will serve as the basis for scientific publication and provide reference data for future development of clinical trials utilizing the endothelin system.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before collection of blood and CSF is commenced.
* TBI diagnosed by history, clinical examination with GCS of 8 or less, and head CT scan and placement of ventriculostomy catheter
* Patients with GCS 9 -12 who undergo placement of a ventriculostomy because of the severity of the CT lesion may be included
* Patients will be enrolled in the study within the first 8 hours after injury
* At least one reactive pupil after injury
* Age 18-70

Exclusion Criteria:

* Life expectancy of less than 8 hours as determined by the investigator
* Associated spinal cord injury
* Patients with penetrating head injury will be excluded
* Inability to establish ventriculostomy drainage
* Severe cardiac or hemodynamic instability consistent with point #1 above
* blood pressure less than 65mmHg mean, will be an exclusion criteria.
* Receipt of any known investigational drug within 30 days prior to this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty patients will be enrolled in this trial. Subjects will be eligible who have severe traumatic brain injury (the majority of patients) or moderate TBI together with lesions on CT scans sufficient to warrant placement of ventriculostomy catheter.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-07; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Ward, MD, Principal Investigator — Virginia Commonwealth University
Locations (11):
- United States (8):
  - University of California, Davis, Sacramento, California
  - Harbor UCLA Medical Center, Torrance, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - The Mayfield Clinic, Cincinnati, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
- University Hospital Heidelberg, Heidelberg, Germany
- University of Padova Medical School, Padua, Italy
- Vall d'Hebron University Hospital, Barcelona, Spain